CLINICAL TRIAL: NCT01822691
Title: A Phase II Study to Determine the Safety and Efficacy of INCB024360 in Patients With Myelodysplastic Syndromes
Brief Title: Phase II INCB024360 Study for Patients With Myelodysplastic Syndromes (MDS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-17280; I-24360-12-01 (Other Grant/Funding Number: Incyte)
Record Dates: First submitted 2013-03-28; First posted 2013-04-02 (Estimated); Results first posted 2016-01-18 (Estimated); Last update posted 2016-01-18 (Estimated); Status verified 2015-11

CONDITIONS: Myelodysplastic Syndromes
Keywords: myelodysplastic syndromes (MDS); neoplastic stem cell disorders; refractory cytopenias; dysplastic morphological features; acute myeloid leukemia (AML)
MeSH Terms: conditions — Myelodysplastic Syndromes; Cytopenia; Leukemia, Myeloid, Acute | interventions — epacadostat; IDO-1 inhibitor LY3381916

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- INCB024360 Treatment (Experimental): Participants were treated with 600 mg orally, twice a day for 16 weeks, unless clear evidence of disease progression or toxicity was evident.
  Interventions: Drug: INCB024360

INTERVENTIONS:
Drug: INCB024360 — INCB024360 is an inhibitor of the enzyme indoleamine 2,3-dioxygenase (IDO) that is proposed for development for the treatment of malignant diseases. Participants were to receive the study drug in 28 day (4 week) cycles of treatment.
  Other Names: inhibitor of indoleamine 2,3-dioxygenase 1 (IDO1); IDO1 inhibitor

SUMMARY:
The primary purpose of this research study is to assess whether the participant's disease, Myelodysplastic Syndromes (MDS), responds favorably to INCB024360. The study will also evaluate the long-term outcomes of the participant's disease after they have finished taking INCB024360.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of myelodysplastic syndromes (MDS)
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
* Adequate organ function:

  * Total bilirubin ≤ 1.5 × Upper Limit of Normal (ULN)
  * Aspartic transaminase (AST)/alanine transaminase (ALT) ≤ 2.5 × ULN
  * Creatinine ≤ 2 × ULN or Creatinine clearance of > 30 mL/min (using the Cockcroft and Gault Equation)
* Females of childbearing potential must have a negative urine or serum pregnancy test at Screening.
* Women of child-bearing potential and men must agree to use adequate contraception (surgical tubal ligation or vasectomy, double-barrier method of birth control condom with spermicide in conjunction with use of an intrauterine device (IUD) or diaphragm; or sexual abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant, or a male impregnate his female partner, while participating in this study, he/she should inform their treating physician immediately.
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Prior MDS therapy within 4 weeks of the first dose of study medication. For erythroid stimulating agent and growth factors: prior therapy with epoetin (Procrit) or G-CSF (neupogen) or GM-CSF (leukine) within 2 weeks of the first dose of study medication.
* Has participated in any other trial in which receipt of an investigational study drug occurred within 28 days.
* Has undergone a stem cell, bone marrow or solid organ transplant.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit by the investigator opinion compliance with study requirements
* History of hepatitis or positive serology as follows:

  * Hepatitis B (HepB) screening testing required: HepB SAg (hepatitis B surface antigen); Anti-HepB SAg (antibody against hepatitis B surface antigen); Anti-Hepatitis B core IgG (antibody against hepatitis B core antigen); Anti-Hepatitis B core IgM antibody Note: Subjects with no prior history of hepatitis B infection who have been vaccinated against hepatitis B and who have a positive anti-HepB SAg test as the only evidence of prior exposure may participate in the trial.
  * Hepatitis C screening required: antibody against hepatitis C virus (HCV-antibody); HCV-RNA (serum test for circulating virus, based on detecting RNA)
* Known history human immunodeficiency virus (HIV)
* Is receiving any compound that is known to be a potent inducer or inhibitor of CYP3A4
* Being treated with a monoamine oxidase inhibitor (MAOI), or drug which has significant monoamine oxidase inhibitory activity (meperidine, linezolid, methylene blue) within 3 weeks prior to screening
* Has, by the investigator assessment, an active autoimmune process such as rheumatoid arthritis, psoriasis, multiple sclerosis, inflammatory bowel disease, etc. or is receiving therapy for an autoimmune disease. Subjects with vitiligo, hypothyroidism or eczema may be enrolled after approval by the sponsor.
* Receiving any immunologically based treatment for any reason, including chronic use of systemic steroid at doses ≥ 7.5 mg/day prednisone equivalents; use of inhaled or topical steroids is acceptable.
* Prior malignancies other than MDS for which the subject has not been disease free for ≤ 3 years, except treated and cured basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the cervix.
* Use of any UGT1A9 inhibitor including: diclofenac, imipramine, ketoconazole, mefenamic acid, and probenecid from screening through follow-up period.
* Have had prior Serotonin Syndrome
* Any unresolved toxicity greater than Grade 2 from previous anticancer therapy, except for stable chronic toxicities not expected to resolve, such as peripheral neurotoxicity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2013-07; Primary Completion 2015-01 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rami Komrokji, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at Moffitt Cancer Center between August 2013 and January 2014.
Period: Overall Study
Arm/Group | INCB024360 Treatment
Started | 15
Completed | 13
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Population: All participants
Arm/Group | INCB024360 Treatment
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 13
Age, Continuous [Median (Full Range); unit: years] | 72 [62 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 12
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: ORR, measured by Response Criteria for Patients with Myelodysplastic Syndrome (MDS). According International Working Group (IWG) 2006 criteria (Cheson et al, 2006). Complete Remission (CR), Partial Remission (PR), Marrow CR, and Hematological Improvement (HI)(any cell line). Stable Disease (SD): Failure to achieve at least PR, but no evidence of progression for > 8 weeks.
Time Frame: Up to 12 months
Population: All participants
Measure: Number; unit: participants
Arm/Group | INCB024360 Treatment
Number analyzed (Participants) | 15
participants
  Stable Disease | 12
  Complete Response | 0
  Marrow Complete Response | 0
  Hematological Improvement | 0
  Progressive Disease | 3

2. Secondary Outcome: Mean Time to Acute Myeloid Leukemia (AML) Progression
Description: Disease progression defined as progression to int-2 or high risk International Prognostic Scoring System (IPSS) score or AML, based on World Health Organization (WHO) AML Criteria.
Time Frame: Up to 12 months
Population: All participants
Measure: Mean (Full Range); unit: months
Arm/Group | INCB024360 Treatment
Number analyzed (Participants) | 15
months | 3.5 [2 to 5]

3. Secondary Outcome: Median Overall Survival (OS)
Description: Overall Survival (OS) defined as the time between the start of treatment and death. Treatment Duration is 17 weeks plus optional continuation phase. Study Duration is Treatment Phase followed by survival follow-up.
Time Frame: Up to 24 months
Population: All participants
Measure: Median (Full Range); unit: months
Arm/Group | INCB024360 Treatment
Number analyzed (Participants) | 15
months | NA [0 to NA] — Median OS was not calculable because an insufficient number of participants reached the event at the final time point for assessment.

4. Secondary Outcome: Number of Participants With Study Related Serious Adverse Events (SAEs)
Description: Participants with treatment emergent Grade 3 or 4 SAEs according to the NCI Common Terminology Criteria for Adverse Events Version (CTCAE) V4.0.
Time Frame: Up to 12 months
Population: All participants
Measure: Number; unit: participants
Arm/Group | INCB024360 Treatment
Number analyzed (Participants) | 15
participants | 0

5. Secondary Outcome: Number of Participants With Study Treatment Related Adverse Events (AEs)
Description: Participants with treatment emergent Other (not including serious) Adverse events.
Time Frame: Up to 12 months
Population: All participants
Measure: Number; unit: participants
Arm/Group | INCB024360 Treatment
Number analyzed (Participants) | 15
participants
  AE of any category | 12
  Metabolism and Nutrition Disorders | 7
  Gastrointestinal Disorders | 6
  General Disorders | 3
  Investigations | 3
  Immune System Disorders | 2
  Musculoskeletal Disorders | 2
  Skin and Subcutaneous Tissue Disorders | 2
  Infections and Infestations | 1
  Nervous System Disorders | 1
  Psychiatric Disorders | 1
  Respiratory Disorders | 1

ADVERSE EVENTS:
Time Frame: 11 months
Arm/Group | INCB024360 Treatment
Serious Adverse Events (participants affected / at risk) | 3/15
Other Adverse Events (participants affected / at risk) | 14/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | INCB024360 Treatment (N=15)
Allergic reaction (Immune system disorders) | 1 (2)
Lung infection (Infections and infestations) | 1 (1)
Lymph gland infection (Infections and infestations) | 1 (1)
Lymphedema (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | INCB024360 Treatment (N=15)
Nausea (Gastrointestinal disorders) | 5 (5)
Constipation (Gastrointestinal disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Oral hemorrhage (Gastrointestinal disorders) | 1 (1)
Platelet count decreased (Investigations) | 4 (8)
Weight loss (Investigations) | 3 (3)
Blood prolactin abnormal (Investigations) | 1 (1)
Investigations - Other, Increased chloride (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 7 (7)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (3)
Metabolism and nutrition disorders - Other, Decreased chloride (Metabolism and nutrition disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, Lip ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Skin induration (Skin and subcutaneous tissue disorders) | 1 (1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1)
Chills (General disorders) | 2 (2)
Fatigue (General disorders) | 2 (2)
Pain (General disorders) | 2 (2)
Irritability (General disorders) | 1 (1)
Upper respiratory infection (Infections and infestations) | 2 (2)
Bladder infection (Infections and infestations) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Immune system disorders - Other, Decreased testosterone (Immune system disorders) | 1 (1)
Immune system disorders - Other, Autoimmune endocrinopathy (Immune system disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (2)
Injury, poisoning and procedural complications - Other, Hand wound (Injury, poisoning and procedural complications) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Confusioin (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1)
Renal and urinary disorders - Other, Kidney injury (Renal and urinary disorders) | 1 (2)

LIMITATIONS AND CAVEATS:
The study was closed prior to meeting the overall survival criteria.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes